CLINICAL TRIAL: NCT04613401
Title: Association of Telemonitoring With Hospitalization Rates and Quality of Life in Patients With End-stage Heart Failure and Implanted Left Ventricular Cardiac Assist Devices
Brief Title: Influence of Telemonitoring on the Management of LVAD-patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Essen (Other)
Responsible Party: Sponsor
Other Study IDs: 20-9312-BO
Record Dates: First submitted 2020-10-26; First posted 2020-11-03 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Heart Failure; Ventricular Assist Device; Telemedicine
MeSH Terms: conditions — Heart Failure | interventions — Surveys and Questionnaires; Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- VAD-patients with Telemonitoring
  Interventions: Other: questionnaire (observational study)

INTERVENTIONS:
Other: questionnaire (observational study) — questionnaire about hospitalisation rates, complications (bleeding, infection, thrombosis), quality of life (Kansas-Score), depression (PHQ8)

SUMMARY:
The current study aims to investigate whether telemedical monitoring in patients with terminal heart failure and an implanted left ventricular assist device (LVAD) has an influence on LVAD-associated complications, hospitalization rates and quality of life. This is a prospective observational study. Patients with terminal heart failure and an implanted LVAD, where the indication for telemonitoring has already been stated by the attending physician are included in the study. Written informed consent is obtained from all patients. The telemedical monitoring is carried out by the West German Center for Applied Telemedicine (WZAT) and includes a standardized telephone interview every 3 days. In addition, all patients are equipped with an INR measuring device, a body scale and a clinical thermometer by WZAT. The data is documented in an electronic case file (medPower®). In the event of abnormalities, the West German Heart and Vascular Center (WHGZ) is contacted, and all necessary measures are initiated.

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years
* Indication for telemedicine
* Permanently implanted left ventricular assist device (VAD)

Exclusion Criteria:

* no possibility of telephone contact
* patient does not speak german
* incompliance
* rejection or inability to give consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with terminal heart failure and LVAD-therapy who are monitored by telemedicine.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Number of days spent in the hospital due to VAD-associated complications | 6 months
  VAD-associated complications are defined as
  * bleeding with the need for a transfusion
  * infection with the need for an antibiotic therapy
  * thrombosis with the need for a lysis therapy

SECONDARY OUTCOMES:
Change in quality of life from baseline | 6 months
  Quality of life will be assessed with the "Kansas City Cardiomyopathy Questionnaire (KCCQ) "
  -> The raw values of the domains are transformed to a scale from 0 to 100, where high values indicate good condition.
Change in depression from baseline | 6 months
  - Depression will be assessed with the "Patient Health Questionnaire eight-item depression scale" (PHQ-8)
  -> The raw values of the domains are transformed to a scale from 0 to 24, where high values indicate a depression.
Number of VAD-associated complications | 6 months
  VAD-associated complications are defined as
  * bleeding with the need for a transfusion
  * infection with the need for an antibiotic therapy
  * thrombosis with the need for a lysis therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Cardiology and Vascular Medicine, West German Heart and Vascular Center, University Hospital Essen, Essen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bundesärztekammer (BÄK) KBK, Arbeitsgemeinschaft der Wissenschaftlichen Medizinischen Fachgesellschaften (AWMF). Nationale VersorgungsLeitlinie Chronische Herzinsuffizienz - Langfassung, 2. Auflage. Version 3. 2017.
- [Background] Bundesauswertung zum Erfassungsjahr 2018: Herzunterstützungssysteme/Kunstherzen; Qualitätsindikatoren und Kennzahlen. IQTIG - Institut für Qualitätssicherung und Transparenz im Gesundheitswesen; 2019 .
- [Result] Reiss N, Schmidt T, Boeckelmann M, Schulte-Eistrup S, Hoffmann JD, Feldmann C, Schmitto JD. Telemonitoring of left-ventricular assist device patients-current status and future challenges. J Thorac Dis. 2018 Jun;10(Suppl 15):S1794-S1801. doi: 10.21037/jtd.2018.01.158. PMID 30034855
- [Result] Kimura M, Nawata K, Kinoshita O, Yamauchi H, Hoshino Y, Hatano M, Amiya E, Kashiwa K, Endo M, Kagami Y, Nemoto M, Ono M. Readmissions after continuous flow left ventricular assist device implantation. J Artif Organs. 2017 Dec;20(4):311-317. doi: 10.1007/s10047-017-0975-4. Epub 2017 Jul 27. PMID 28752193
- [Result] Smedira NG, Hoercher KJ, Lima B, Mountis MM, Starling RC, Thuita L, Schmuhl DM, Blackstone EH. Unplanned hospital readmissions after HeartMate II implantation: frequency, risk factors, and impact on resource use and survival. JACC Heart Fail. 2013 Feb;1(1):31-9. doi: 10.1016/j.jchf.2012.11.001. Epub 2013 Feb 4. PMID 24621797
- [Result] Reiss N, Wegner KK, Hoffmann JD, Schulte Eistrup S, Boeken U, Morshuis M, Schmidt T. Requirements for a Telemedicine Center to Monitor LVAD Patients. Stud Health Technol Inform. 2019;260:146-153. PMID 31118331
- [Result] Bohm M, Drexler H, Oswald H, Rybak K, Bosch R, Butter C, Klein G, Gerritse B, Monteiro J, Israel C, Bimmel D, Kaab S, Huegl B, Brachmann J; OptiLink HF Study Investigators. Fluid status telemedicine alerts for heart failure: a randomized controlled trial. Eur Heart J. 2016 Nov 1;37(41):3154-3163. doi: 10.1093/eurheartj/ehw099. Epub 2016 Mar 16. PMID 26984864
- [Result] Hindricks G, Taborsky M, Glikson M, Heinrich U, Schumacher B, Katz A, Brachmann J, Lewalter T, Goette A, Block M, Kautzner J, Sack S, Husser D, Piorkowski C, Sogaard P; IN-TIME study group*. Implant-based multiparameter telemonitoring of patients with heart failure (IN-TIME): a randomised controlled trial. Lancet. 2014 Aug 16;384(9943):583-590. doi: 10.1016/S0140-6736(14)61176-4. PMID 25131977
- [Result] Koehler F, Koehler K, Deckwart O, Prescher S, Wegscheider K, Kirwan BA, Winkler S, Vettorazzi E, Bruch L, Oeff M, Zugck C, Doerr G, Naegele H, Stork S, Butter C, Sechtem U, Angermann C, Gola G, Prondzinsky R, Edelmann F, Spethmann S, Schellong SM, Schulze PC, Bauersachs J, Wellge B, Schoebel C, Tajsic M, Dreger H, Anker SD, Stangl K. Efficacy of telemedical interventional management in patients with heart failure (TIM-HF2): a randomised, controlled, parallel-group, unmasked trial. Lancet. 2018 Sep 22;392(10152):1047-1057. doi: 10.1016/S0140-6736(18)31880-4. Epub 2018 Aug 25. PMID 30153985
- [Result] Berg T, Tewarie L, Moza A, Zayat R, Autschbach R, Stoppe C, Goetzenich A, Benstoem C. [Requirements for outpatient care after implantation of a ventricular assist device : Views of patients and their relatives]. Herz. 2019 May;44(3):257-264. doi: 10.1007/s00059-017-4636-4. Epub 2017 Oct 27. German. PMID 29079934